CLINICAL TRIAL: NCT03951870
Title: Characterization of the Relationship Between the Mesolimbic Reward System and Immune Functioning in Humans Via fMRI Neurofeedback
Brief Title: Characterization of the Relationship Between the Human Mesolimbic Reward System and Immune Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0664-17-TLV
Record Dates: First submitted 2019-04-17; First posted 2019-05-15 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-07

CONDITIONS: Immune Hepatitis
Keywords: mesolimbic reward system; fMRI Neurofeedback

STUDY DESIGN:
Intervention Model Description: 1. Experimental arm: fMRI neurofeedback to mesolimbic system (the ventral tegmental area, and bilateral ventral striatum).
  2. Active control arm: fMRI neurofeedback to a control network.
  3. Natural history arm: assessment of immunological response to Hepatitis B without neurofeedback manipulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both participants and study personnel (Investigators and outcomes assessor) in the two active experimental arms (Mesolimbic NF and Control NF) will be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mesolimbic Neurofeedback (Experimental): Neuromodulation via fMRI Neurofeedback task: subjects (n=34) will participate in four fMRI-NF sessions, up-regulating activation of three mesolimbic reward nodes:
  ventral tegmental area, and bilateral ventral striatum. ROIs are 5 mm spheres around peak activations in funcitonal localizer task (Monetary Incentive delay, reward anticipation contrast), within a predifned meta-analytic anatomical masks of the three regions.
  anatomical masks: VTA (Midbrain): -4 -24 -10 *see below Right Nac: 12 10 -4 Left Nac: -10 10 -6 Oldham, Stuart, et al. Human brain mapping (2018).
  * 23/08/22: Due to VTA complex contours, it was not restricted according to Oldham et al as mentioned above, but via more accurate VTA mask (Murty et al. 2014, NeuroImage). This was mistakenly left out of the original preregistration. It is noteworthy that, to date (23/8/22), ROI analyses haven't been performed.
  Hepatitis B vaccination: subjects will receive vaccination against Hepatitis B.
  Interventions: Behavioral: Neuromodulation via fMRI Neurofeedback task; Biological: Hepatitis B vaccination
- Control Neurofeedback (Active Comparator): Neuromodulation via fMRI Neurofeedback task: subjects (n=34) will participate in four fMRI-NF sessions, up-regulating activation of regions comprising one of 4 control networks (5mm spheres around MNI coordinates):
  Motor Imagery (Hétu, Sébastien, et al. Neurosci. & Biobehav Rev (2013)) R. Cerebellum: 32 -62 -28 L. Cerebellum: -32 -56 -30 L. Precentral Gyrus: -26 -2 58; Auditory imagery (McNorgan, Chris.Front in Human Neurosci 6 (2012)) R STG:64 -30 9 L IFG:-48 24 -5 L precentral Gyrus: -52 1 47; Arithmetic processing (Arsalidou, Marie, and Margot J. Taylor. Nuroimage (2011)) R. SPL: 29 -66 49 L. MFG (dlpfc): -45 32 29 L. precuneus: -28 -71 33; Spatial Navigation (Kühn, Simone, and Jürgen Gallinat. Human Brain Map. (2014)) R. hippocampus 26 -35 -11 L. hippocampus -26 -47 -9 L. Post. cingulate -15 -59 19
  Hepatitis B vaccination: subjects will receive vaccination against Hepatitis B.
  Interventions: Behavioral: Neuromodulation via fMRI Neurofeedback task; Biological: Hepatitis B vaccination
- Natural history (Other): No brain manipulation (Assesment of natural history immune response).
  Hepatitis B vaccination: subjects (n=17) will receive vaccination against Hepatitis B.
  Interventions: Biological: Hepatitis B vaccination

INTERVENTIONS:
Behavioral: Neuromodulation via fMRI Neurofeedback task — Two active neurofeedback groups will practice to up regulate their designated neural targets via identical experimental protocol (varying only the origin of the feedback).
  Arms: Control Neurofeedback; Mesolimbic Neurofeedback
Biological: Hepatitis B vaccination — Subjects will be vaccinated against Hepatitis B

SUMMARY:
The purpose of this study is to characterize the link between neurobehavioral measures of the mesolimbic reward system and immune functioning in healthy individuals, via fMRI neurofeedback modulation of mesolimbic reward system, and the consecutive assesment of immune response to Hepatitis B vaccination.

DETAILED DESCRIPTION:
For many years, the link between mental processes and physical health has remained obscure. Yet, over time, studies have begun to shed light on the intimate relationship between one's physical condition and mental state. One body of research aimed at elucidating the mind-body relationship is the study of the placebo effect. Placebo effects result mainly from conscious expectations to become healthy in therapeutic settings, and from unconscious conditioned responses to therapeutical settings that predict beneficial outcomes. Both processes are asociated with the neuronal reward system, which mediates reward processing, reward valuation and value based-learning. However, it remains unclear how do these processes mediated by the reward system promote therapeutic effects?

A recent study established a causal relationship between mesolimbic activation (VTA) and a measurable immunological response in mice. Stimulation of the VTA increased anti-bacterial immune functioning, an effect that was mediated by sympathetic nervous system, which is regulated by the brain and innervates all immune organs.

In light of these findings, the current study aims to assess the relationship between reward-related brain activation and immune functions in humans. fMRI Neurofeedback, a task that allows individuals to self modulate specified neural patterns in real-time, will be used to induce mesolimbic activation, following which healthy individuals will vaccinate against Hepatitis B. Immunological effects will be assessed by comparing immunological measures with respect to Hepatitis B prior and following mesolimbic activation and Hepatitis B vaccination.

The long-term goal of this study is to demonstrate a causal link between reward activation and an objective measurable physiological response of great significance, and to develop the means for individuals to exploit such mechanism for boosting immune functioning. i.e. to harness endogenous reward-related brain activation to strengthen the immune system, for clinical pathologies such as autoimmune diseases, maleble pathogens, cancer, etc.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Normal or corrected to normal vision
* Compatibility with general MRI requirements

Exclusion Criteria:

* History of neurological or psychiatric diseases that lead to hospitalization
* Have received Hepatitis B vaccination in the last 10 years
* Memory/cognitive neurological impairments
* Chronic heart disease, diabities, high blood pressure, or autoimmune disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Immunological: change in anti HBs immunoglobins in plasma | 6 weeks
  To measure antibody titers in plasma, blood samples will be taken at four time points: before neurofeedback training (-14d); before Hepatitis B vaccination (day 0), 14 days and 28 days after vaccination. Anti-HBs change will be defined as average levels post-vaccination (14 and 28 days) minus average levels pre-vaccination (-14 and 0 days).
  *19.09.22: due to extensive variability in baseline levels, anti-HB change will be defined as fold change between pre-and post-vaccination TPs, instead of absolute differences (blinding unharmed).
  The investigators predict that:
  i.Simple group effect: experimental arm subjects (mesolimbic fMRI NF) will exhibit higher levels of anti-HBs change than both the active comparator group (control fMRI-NF) and the no-treatment group.
  ii.Mesolimbic activation-Immunologic response correlation: mesolimbic activity during the neurofeedback task (across all NF participants) during the last session will predict anti-HBs levels following vaccination.
Immunological: change in cytokines blood concentrations following vaccination | 17 days
  To assess cytokine levels (e.g. IL-4, IL-6, TNFalpha, IFNgamma), the investigators will isolate peripheral blood mononuclear cells from the blood, and using flow cytometry analysis, characterize cytokine expression profile (initial intentions of using ELISA will be replaced due to quality tests (blinding unharmed) that showed poor signal, 28/12/21). As mere NF practice may affect cytokines levels, cytokines will be assessed in three time points - before NF training (-14d), before vaccination (day 0) and 3 days following vaccination. groupXtime (3X3) main effect and interactions will be inspected.
  The investigators predict that:
  i.Experimental arm group will exhibit higher levels of cytokines concentration that the active control group and natural history group.
  ii.Mesolimbic activation-Immunologic response correlation: mesolimbic activity during the neurofeedback task (across all NF participants) during the last session will predict changes in cytokines blood concentrations.
Reward Mesolimbic network (or control networks) BOLD activity during fMRI-NF task | 1-3 weeks
  ROIs of Mesolimbic reward network (or control networks) will be defined as mentioned in arms description *see below. CSF voxels will be excluded from all ROIs. Outcome will be measured for each experimental group/control sub-group, as the contrast between regulation and watch conditions, for each NF run, each session (3*4=12 runs).
  To assess differences in meoslimbic reward network activation between experimental and active control groups, a 12 by 2 (runXgroup) model will be constructed.
  *23/8/22 to exploit superior offline processing, ROIs will be deifned via group instead of online individual subs analysis.
  The investigators predict that:
  i. Simple group effects during last (fourth) NF session: experimental arm subjects (mesolimbic fMRI NF) will exhibit higher meoslimbic reward network activity than the active comparator group.
  ii. Simple experimental arm group learning effects: a significant effect of run (time) for the experimental arm mesolimbic reward network acitivity.

SECONDARY OUTCOMES:
Mental Strategies Questionnaire for NeuroFeedback (MSQ-NF) | 6 weeks
  For each NF cycle in their training, subjects will fill out the MSQ-NF, a quesitonnaire that characterize mental strategies according to a hierarchical mental categorization.
  Exploratory analysis: The investigators suspect that mental features that relate to motivation and reward processing will be associated with reward mesolimbic activity during NF training, and that such mental features will be associated post-practice immunological effects.
Neurobehavioral measures of reward anticipation and responsivity during Monetary Incentive Delay (MID) task. | 6 weeks
  Neurobehavioral measures of reward responsitivity and reward anticipation will be assessed via application of MID task during fMRI scanning at the beginning of the first fMRI session (for all three study groups).
  The investigators intend to explore whether neural and behavioral indices of reward anticipation and consumption could account for differences in immunological outcome measures, as defined above (see primary outcome measures).
  Specifically, the investigators predict that:
  i. BOLD responses to reward anticipation will be positively correlated with immunological outcome measures - Cytokines levels change and HBV antibodeis change (as defined above).
Behavioral measures of incentive motivation extracted from Effort Expenditure for Rewards Task (EEfRT). | 6 weeks
  Behavioral measures of incentive saliance and incentive motivation will be assessed via application of EEfRT at the beginning of the first experimental session (for all three study groups).
  The investigators intend to explore whether EEfRT scores could account for differences in immunological and NF success outcome measures, as defined above (see primary outcome measures).
Motivational tendencies based on K-means cluster analysis of questionnaires scores | 6 week
  Subjects' classification as having approach/avoidance tendencies based on K-means cluster analysis of scores in three questionnaires: SPSRQ, TPQ and NEO-ffi.
  The investigators predict that:
  i. subjects with approach tendencies will exhibit stronger mesolimbic reward network activations during the MID task and NF task, compared to avoiders.
  ii. Approachers will exhibit higher immunological changes as reflected by the main immunological outcome measures, compared to avoiders.
Functional connectivity of mesolimbic network during rest fMRI scan | 1-3 weeks
  Rest scans will be applied at the beginning of the first and at the end of the fourth (last) NF practice session, in order to assess functional changes in the mesolimbic reward circuit following NF training.
  The investigators intend to explore whether changes in functional connectivity of the mesolimbic reward network will occur specifically in the mesolimbic fMRI-NF group (compared with control fMRI NF group).
long term immunological effects | 3 months
  A sub-group of 30 subjects will arrive for an aditional blood sample session three months following vaccination, in order to assess long term differences in anti-HBs levels.
  Exploratory analysis: differences between groups and brain-immune correlations will be examined.
Subjective reports of SHAPS (Snaith-Hamilton Pleasure Scale) | 6 weeks
  A 14 items (answered on a four points scale ranging from 'strongly disagree' to 'strongly agree') questionnaire for estimation of the degree of which a person is able to experience pleasure or the anticipation of a pleasurable experience. The questionnaire is scored as the sum of of the items (totals scores ranged from 0 to 14). A higher total score indicates higher levels of anhedonia.
  Exploratory Analyses: The investigators will examine whether the questionnaire scores prior to NF practice and vaccination, will account for differences in NF learning and in immunological outcome measures. Moreover, the investigators will track changes in this score along the experiment in order to inspect the relationship between subjective hedonic experience and NF success/immune functioning.
Subjective reports to Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) | 6 weeks
  A questionnaire for assessing responsiveness to reward and punishment. The questionnaire includes 48 yes/no questions divided into two scales - sensitivity to punishment (SP) and sensitivity to reward (SR). Each sub-scale score is derived by summation of the reports.
  Exploratory analysis: the investigators will examine whether the questionnaire score during the first session (prior to NF practice and vaccination), will account for differences in NF learning and in immunological outcome measures.
Subjective reports to Tridimensional Personality Questionnaire (TPQ) | 6 weeks
  A questionnaire with 100 true/false items to characterize individual's three traits of personality - reward dependence, harm avoidance and novelty seeking. Each trait has 4 sub-scales that sums to the trait's score.
  Exploratory analysis: the investigators will examine whether the questionnaire score during the first session (prior to NF practice and vaccination), will account for differences in NF learning and in immunological outcome measures.
Autonomic Nervous System (ANS) measure: Heart Rate Variability (HRV) | 3 days - 4 weeks
  Measurements of HRV are taken during fMRI scans in all NF practices, in order to monitor the activity of the sympathetic system. For each fMRI scan, HRV measures such as average variability and frequency ratios will be calculated.
  Exploratory analyses: the investigators suspect the sympathetic system will mediate the correlation between the mesolimbic reward activations and immunological outcome meaures (see primary outcome measures 1 and 2). Therefore, the investigators will explore the link between sympathetic measures taken at TP4 (prior to vaccination) and the correlation between reward mesolimbic activations during TP4 NF practice and the immunological outcome measures described above.

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, MD, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Functional Brain Center, Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lubianiker N, Koren T, Djerasi M, Sirotkin M, Singer N, Jalon I, Lerner A, Sar-El R, Sharon H, Shahar M, Azulay-Debby H, Rolls A, Hendler T. Upregulation of reward mesolimbic activity and immune response to vaccination: a randomized controlled trial. Nat Med. 2026 Jan 19. doi: 10.1038/s41591-025-04140-5. Online ahead of print. PMID 41555034